CLINICAL TRIAL: NCT03603977
Title: A Simplified Therapy Regimen Study of Lopinavir and Ritonavir Combined With Lamivudine for HIV-1 Infected Patients in the Real World of China
Brief Title: Simplified Treatment of Anti-retrovirus in China (C-STAR)
Status: Recruiting | Type: Observational
Sponsor: Guangzhou 8th People's Hospital (Other)
Collaborators: Guiyang Public Health Clinical Center (Unknown); The Third People's Hospital of Kunming (Unknown); The Second People's Hospital of Nanjing (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Third People's Hospital of Guilin (Unknown); Guangxi Longtan hospital (Unknown); The Fourth People's Hospital of Nanning (Other); LiuZhou People's Hospital (Other); Tianjin Second People's Hospital (Other); The Sixth People's Hospital of Shenyang (Other); The Sixth People's Hospital of Henan (Unknown); The Sixth People's Hospital of Xinjiang (Unknown); The Eighth People's Hospital of Xi'an (Unknown)
Responsible Party: Principal Investigator, Linghua LI, Vice Chief physician, Guangzhou 8th People's Hospital
Other Study IDs: GZ8H-2017014
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: HIV/AIDS
Keywords: Simplified Therapy Regimen; Real World Study; HIV-1-infected patients
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lpv/r+3TC: These cases were given simplified therapy regimen including lopinavir(200mg) and ritonavir(50mg)500 mg,oral,bid) combined with lamivudine (300 mg,oral,qd).
  Interventions: Drug: Lpv/r+3TC

INTERVENTIONS:
Drug: Lpv/r+3TC — It is a simplified therapy regimen study of lopinavir and ritonavir combined with lamivudine for HIV-1 infected patients in the real world of China.
  Other Names: A simplified therapy regimen

SUMMARY:
To observe the efficacy and safety of simplified therapy regimen for treating with HIV-1 infected patients in Chinese real word.

DETAILED DESCRIPTION:
This is an phase IV open-label, multicenter, single-arm clinical trial in. A total of 600 cases were planned to be recruited. These cases were given simplified therapy regimen of lopinavir (200mg) and ritonavir (50mg) (500mg, oral, bid ) combined with lamivudine (300mg, oral, qd. The observation duration is thirty-sixth months. Patients will be followed up before and 12, 24 and 36 months after receiving the simplified regimen, observing the viral inhibition rate and the change of CD4 cell count, the safety and patients'compliance.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection confirmed
2. Agree to use simplified therapy regimen.
3. Agree to detect CD4 count at least once per half a year

Exclusion Criteria:

1. Have participated in HIV vaccine clinical trial or other drug trials in the past three months.
2. Patients who could not complete the scheduled follow-up (such as weakness and poor compliance).
3. Patients who have the history of resistance or allergy to LPV/r or 3TC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are prescribed to take the simplified therapy regimen (LPV/r+ 3TC) because they are unable to tolerate the side-effect of or are not fit for the first-line free regimen in China, for example renal failure or osteoporosis, according to clinical judgment, no matter of the HIV-RNA viral loads and CD4 cell counts.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
The rate of virus inhibition | 36 Months
  the ratio of HIV RNA< 50 copies/mL at 12, 24 or 36 months after treatment.

SECONDARY OUTCOMES:
The immunological ability | 36 Months
  the count of CD4 cells

OTHER OUTCOMES:
The level of compliance | 36 Months
  To explicit the number of people who have completed the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Cai, Bachelor, Study Chair — Guangzhou 8th People's Hospital
Locations (1):
- Guangzhou 8th People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cahn P, Andrade-Villanueva J, Arribas JR, Gatell JM, Lama JR, Norton M, Patterson P, Sierra Madero J, Sued O, Figueroa MI, Rolon MJ; GARDEL Study Group. Dual therapy with lopinavir and ritonavir plus lamivudine versus triple therapy with lopinavir and ritonavir plus two nucleoside reverse transcriptase inhibitors in antiretroviral-therapy-naive adults with HIV-1 infection: 48 week results of the randomised, open label, non-inferiority GARDEL trial. Lancet Infect Dis. 2014 Jul;14(7):572-80. doi: 10.1016/S1473-3099(14)70736-4. Epub 2014 Apr 27. PMID 24783988
- [Background] Arribas JR, Girard PM, Landman R, Pich J, Mallolas J, Martinez-Rebollar M, Zamora FX, Estrada V, Crespo M, Podzamczer D, Portilla J, Dronda F, Iribarren JA, Domingo P, Pulido F, Montero M, Knobel H, Cabie A, Weiss L, Gatell JM; OLE/RIS-EST13 Study Group. Dual treatment with lopinavir-ritonavir plus lamivudine versus triple treatment with lopinavir-ritonavir plus lamivudine or emtricitabine and a second nucleos(t)ide reverse transcriptase inhibitor for maintenance of HIV-1 viral suppression (OLE): a randomised, open-label, non-inferiority trial. Lancet Infect Dis. 2015 Jul;15(7):785-92. doi: 10.1016/S1473-3099(15)00096-1. Epub 2015 Jun 7. Erratum In: Lancet Infect Dis. 2015 Aug;15(8):875. doi: 10.1016/S1473-3099(15)00112-7. PMID 26062880
- [Background] Ciaffi L, Koulla-Shiro S, Sawadogo AB, Ndour CT, Eymard-Duvernay S, Mbouyap PR, Ayangma L, Zoungrana J, Gueye NFN, Diallo M, Izard S, Bado G, Kane CT, Aghokeng AF, Peeters M, Girard PM, Le Moing V, Reynes J, Delaporte E; MOBIDIP study group. Boosted protease inhibitor monotherapy versus boosted protease inhibitor plus lamivudine dual therapy as second-line maintenance treatment for HIV-1-infected patients in sub-Saharan Africa (ANRS12 286/MOBIDIP): a multicentre, randomised, parallel, open-label, superiority trial. Lancet HIV. 2017 Sep;4(9):e384-e392. doi: 10.1016/S2352-3018(17)30069-3. Epub 2017 May 28. PMID 28566227